CLINICAL TRIAL: NCT05163223
Title: A Phase 2 Study to Evaluate the Efficacy and Safety of an Adjuvant Therapeutic Cancer Vaccine (AST-301, pNGVL3-hICD) in Patients With HER2 Low Breast Cancer (Cornerstone-001)
Brief Title: Therapeutic Cancer Vaccine (AST-301, pNGVL3-hICD) in Patients With Breast Cancer
Acronym: Cornerstone001
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in recruiting patients
Sponsor: Aston Sci. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PN-301-21
Record Dates: First submitted 2021-04-02; First posted 2021-12-20 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
Keywords: HER 2 low (1+ or 2+ and non-amplified by FISH)
MeSH Terms: conditions — Breast Neoplasms | interventions — sargramostim; Saline Solution; pembrolizumab; Capecitabine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AST-301(pNGVL3-hICD)+Chemotherapy (Experimental): * AST-301/rhuGM-CSF (q 3 weeks, 3 cycles) + Standard adjuvant therapy*
  * A booster (AST-301/rhuGM-CSF) at 24 weeks post the third vaccination
    * Standard adjuvant therapy will be pembrolizumab or capecitabine (q 3 weeks)
  Interventions: Biological: AST-301(pNGVL3-hICD); Drug: rhuGM-CSF; Drug: Pembrolizumab; Drug: Capecitabine
- Placebo + Chemotherapy (Active Comparator): * Placebo/rhuGM-CSF (q 3 weeks, 3 cycles) + Standard adjuvant therapy*
  * A booster (Placebo/rhuGM CSF) at 24 weeks post the third vaccination
    * Standard adjuvant therapy will be pembrolizumab or capecitabine (q 3 weeks)
  Interventions: Drug: rhuGM-CSF; Drug: Placebo; Drug: Pembrolizumab; Drug: Capecitabine

INTERVENTIONS:
Biological: AST-301(pNGVL3-hICD) — Q3W, 3 cycles, Plus a booster at 24 weeks post the third vaccination, Intradermal injection
  Other Names: AST-301
  Arms: AST-301(pNGVL3-hICD)+Chemotherapy
Drug: rhuGM-CSF — Q3W, 3 cycles, Plus a booster at 24weeks post the third vaccination, Intradermal injection
  Other Names: Leukine; Sargramostim
Drug: Placebo — Q3W, 3 cycles, Plus a booster at 24 weeks post the third vaccination, Intradermal injection
  Other Names: Normal Saline
  Arms: Placebo + Chemotherapy
Drug: Pembrolizumab — Q3W; IV infusion
  Other Names: Keytruda
Drug: Capecitabine — On days 1-14 (Q3W), BID ; Oral administration,
  Other Names: Xeloda

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of an adjuvant treatment of therapeutic cancer vaccine (AST-301, pNGVL3-hICD) in patients with HER2-low expression (IHC 1+ or 2+ and ISH-) and hormone receptor-negative(ER-, PR-) breast cancer with residual disease after neoadjuvant treatment.

Patients will be randomized 1:1 to either the Experimental arm (combination of AST-301/rhuGM CSF and standard adjuvant therapy) or the Control arm (combination of placebo/rhuGM CSF and standard adjuvant therapy). Standard adjuvant chemotherapy will be pembrolizumab or capecitabine.

Adjuvant therapy will be administered in compliance with the NCCN guideline for breast cancer (Version 8, 2021), and IP (AST-301) will be administered 3 times every 3 weeks in the adjuvant treatment period, with a booster administered at 24 weeks (±7 days) post the third dose of IP administration.

Survival follow up will be performed to determine invasive Disease Free survival(iDFS).

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Key Inclusion Criteria:

* Has a residual invasive cancer in the breast(non-pCR) after neoadjuvant treatment
* Has stage I, II, or III disease prior to surgery per American Joint Committee on Cancer (AJCC)
* HER 2 1+ by IHC or HER2 2+by IHC without gene amplification by ISH, as defined by American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines.
* Hormone receptor (ER and PR) negative by ASCO/CAP guidelines
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Demonstrates adequate organ function.

Key Exclusion Criteria:

* Has a history of hypersensitivity or other contraindications to rhGM-CSF
* Has a history of invasive malignancy ≤5 years prior to first administration of investigational drug except for adequately treated non-melanoma skin cancer or carcinoma in situ.
* Is on immune suppression therapy or has a history of immune suppression therapy ≤4 weeks prior to the first administration of investigational drugs
* Has a history of autoimmune disease or inflammatory disease
* Has active infection including tuberculosis, hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection
* Is pregnant or breastfeeding or expecting to conceive children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
2-year invasive disease free survival rate (iDFS) | Overall study period approximately up to 4years (End of study in this study is defined as 2years frm the date of last Patient In.
  iDFS event is defined as Ipsilateral breast tumor recurrence Local/regional invasive recurrence Distant recurrence Invasive contralateral breast cancer Death (from breast cancer/non-breast cancer cause/unknown cause) Secondary primary invasive cancer (non-breast)

SECONDARY OUTCOMES:
AST-301 specific T cell immune responses | Up to approximately 82 weeks
  Immune response will be assessed by IFN-gamma enzyme-linked immune absorbent spot (ELISpot) assay
Change in central memory T cell populations | Up to approximately 82 weeks
  Assessment by FACS
Distant Recurrence-Free Survival rate, dRFS rate | Overall study period approximately up to 4 years
  dRFS rate at the end of study
Number of participants with treatment-related adverse events as assessed by CTCAE | Overall study period approximately up to 4years
  To assess safety of AST-301 administered in breast cancer patients.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (10):
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - Scripps Health, La Jolla, California
  - Moffitt Cancer Center, Tampa, Florida
  - University of Illinois Cancer Center, Chicago, Illinois
  - Nebraska Cancer Specialist, Omaha, Nebraska
  - Gabrail Cancer Center Research, Canton, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Providence Cancer Institute, Portland, Oregon
  - University of Washington, Seattle, Washington
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chi Mei Medical Center, Tainan
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No